CLINICAL TRIAL: NCT02954341
Title: CardioMEMS HF System OUS Post Market Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10147
Record Dates: First submitted 2016-10-21; First posted 2016-11-03 (Estimated); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Left-Sided Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CardioMEMS HF System

SUMMARY:
The purpose of this Post Market Study (PMS) is to evaluate the use of the CardioMEMS HF System in patients with New York Heart Association (NYHA) Class III Heart Failure in a commercial setting.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from subject
2. ≥ 18 years of age
3. Diagnosis of NYHA Class III Heart Failure
4. At least 1 HF hospitalization within 12 months of Baseline visit
5. Subjects with reduced LVEF heart failure should be receiving a beta blocker for 3 months and an ACE-I or ARB for one month unless in the investigator's opinion, the subject is intolerant to beta blockers, ACE-I or ARB.
6. Subjects with a BMI ≤ 35. Subjects with BMI >35 will require their chest circumference to be measured at the axillary level, if > 65 inches the patient will not be eligible for the study.
7. Subjects with pulmonary artery branch diameter ≥ 7mm - (implant target artery - assessed during the RHC)
8. Subjects willing and able to comply with the follow-up requirements of the study

Exclusion Criteria:

1. Subjects with an active infection
2. Subjects with history of recurrent (> 1) pulmonary embolism or deep vein thrombosis
3. Subjects who, in the Investigator's opinion, are unable to tolerate a right heart catheterization
4. Subjects who have had a major cardiovascular event (e.g., myocardial infarction, open heart surgery, stroke, etc.) within 2 months of Baseline Visit
5. Subjects with Cardiac Resynchronization Device (CRT) implanted < 3 months prior to enrollment
6. Subjects with a Glomerular Filtration Rate (GFR) < 25 ml/min (obtained within 2 weeks of the baseline visit) who are non-responsive to diuretic therapy or who are on chronic renal dialysis
7. Subjects with congenital heart disease or mechanical right heart valve(s)
8. Subjects likely to undergo heart transplantation or VAD within 6 months of baseline visit
9. Subjects with known coagulation disorders
10. Subjects with a hypersensitivity or allergy to aspirin, and/or clopidogrel (not applicable for subjects taking anti-coagulation therapy or other approved anti-platelets therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with New York Heart Association (NYHA) Class III Heart Failure (HF) who have experienced a heart failure hospitalization within the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal De Groote, MD, Study Chair — CHU de Lille - Institut Coeur Poumon
Locations (5):
- The Prince Charles Hospital, Chermside, Queensland, Australia
- CHR Citadelle, Liège, Belgium
- Rigshospitalet, Copenhagen, Denmark
- CHRU de Lille, Lille, France
- Royal Bromptom Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cowie MR, Flett A, Cowburn P, Foley P, Chandrasekaran B, Loke I, Critoph C, Gardner RS, Guha K, Betts TR, Carr-White G, Zaidi A, Lim HS, Hayward C, Patwala A, Rogers D, Pettit S, Gazzola C, Henderson J, Adamson PB. Real-world evidence in a national health service: results of the UK CardioMEMS HF System Post-Market Study. ESC Heart Fail. 2022 Feb;9(1):48-56. doi: 10.1002/ehf2.13748. Epub 2021 Dec 9. PMID 34882989
- [Derived] Cowie MR, de Groote P, McKenzie S, Brett ME, Adamson PB; CardioMEMS Post-Market Study Investigators. Rationale and design of the CardioMEMS Post-Market Multinational Clinical Study: COAST. ESC Heart Fail. 2020 Jun;7(3):865-872. doi: 10.1002/ehf2.12646. Epub 2020 Feb 7. PMID 32031758

RESULTS

PARTICIPANT FLOW:
Groups:
- Consented Population: Patients who signed the study Informed Consent
Period: Overall Study
Arm/Group | Consented Population
Started | 321
Underwent Implant (Safety Population) | 304
Successfully Implanted (Effectiveness Population) | 299
Completed | 190
Not Completed | 131
Not completed — Attempted Implant unsuccessful | 5
Not completed — Death | 90
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 13
Not completed — Not Implanted due to COVID restrictions | 1
Not completed — Not implanted due to physician's decision | 1
Not completed — Withdrawn Prior Implant Attempt | 17

BASELINE CHARACTERISTICS:
Population: Patients who underwent a successful implant constitute the Effectiveness Population
Groups:
- Effectiveness Population: Patients who signed the Study Informed Consent and underwent successful CardioMEMS implant
Arm/Group | Effectiveness Population
Number analyzed (Participants) | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 218
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Ischemic Cardiomyopathy [Count of Participants; unit: Participants] — Patients with Ischemic Cardiomyopathy
  Participants | 137
CRT/CRT-D [Count of Participants; unit: Participants] — Patients with Cardiac Resynchronization Therapy (CRT) or Cardiac Resynchronization Therapy with Defibrillation (CRT-D)
  Participants | 87
ICD [Count of Participants; unit: Participants] — Patients with Implantable Cardioverter Defibrillator (ICD)
  Participants | 71
Preserved Ejection Fraction (EF) [Count of Participants; unit: Participants] — Patients with Ejection Fraction higher than 40% at baseline
  Participants | 106
Hypertension [Count of Participants; unit: Participants] — Patients diagnosed with hypertension at baseline
  Participants | 164
Diabetes Mellitus [Count of Participants; unit: Participants] — Patients diagnosed with Diabetes Mellitus at baseline
  Participants | 129
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] — Patients diagnosed with Chronic obstructive pulmonary disease at baseline
  Participants | 67
Chronic kidney disease [Count of Participants; unit: Participants] — Patients diagnosed with Chronic kidney disease at baseline are then categorized in stages (1 to 5) depending on the estimated Glomerular Filtration Rate (eGFR), Stage 1 is less serious than stage 5:
  stage 1: a normal eGFR above 90ml/min, but other tests have detected signs of kidney damage stage 2: a slightly reduced eGFR of 60 to 89ml/min, with other signs of kidney damage stage 3: an eGFR of 30 to 59ml/min stage 4:an eGFR of 15 to 29ml/min stage 5:an eGFR below 15ml/min, meaning the kidneys have lost almost all of their function Population: Only Chronic Kidney disease of stage 3, 4 and 5 were collected therefore if a patient had a CKD in stage 2, it was not reported.
  Participants
    Stage 3 | 187
    Stage 4 | 23
    Stage 5 | 1
    Not collected/Not reported | 88
Glomerular filtration rate (eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Glomerular filtration rate (mL/min/1.73 m2) measured at baseline
  mL/min/1.73 m^2 | 51.53 (19.85)
Medications at baseline [Number; unit: number of patients taking medication] — Patient medications at baseline
  number of patients taking medication
    Beta Blockers | 248
    ACE inhibitor/ARB/ARNi | 255
    Beta Blocker + ACE inhibitor/ARB/ARNi | 202
    Mineralocorticoid Receptor Antagonists (MRA) | 66
    Diuretics (all types) | 293
    Loop Diuretic | 288
    Thiazide Diuretic | 47
    Other diuretics | 133
NYHA Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional class helps to classify congestive heart failure patients based on their symptoms. Its classes are:
  Class I: No symptoms of heart failure. Class II: Symptoms of heart failure with moderate exertion, such as ambulating two blocks or two flights of stairs.
  Class III: Symptoms of heart failure with minimal exertion, such as ambulating one block or one flight of stairs, but no symptoms at rest.
  Class IV: Symptoms of heart failure at rest.
  Participants
    Class I | 0
    Class II | 0
    Class III | 299
    Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Device/System Related Complications
Description: A device/System related complication (DSRC) is an adverse event that is, or is possibly, related to the device/system (wireless pressure sensor or external electronics) and has at least one of the following characteristics: 1) is treated with invasive means (other than intramuscular medication or right heart catheterization which is used for diagnostic purposes); 2) results in death of the subject; 3) results in the explant of the device.
Time Frame: Two year
Population: Patients who signed the study Informed Consent and underwent CardioMEMS implant
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: Patients who signed the study Informed Consent and underwent CardioMEMS implant procedure
Arm/Group | Safety Population
Number analyzed (Participants) | 304
Participants | 304

2. Primary Outcome: Freedom From Pressure Sensor Failure.
Description: A sensor failure occurs when no readings can be obtained from it after troubleshooting the system to rule out any problems with the external electronics.
Time Frame: Two year
Measure: Count of Participants; unit: Participants
Arm/Group | Effectiveness Population
Number analyzed (Participants) | 299
Participants | 298

3. Primary Outcome: Annualized Heart Failure Hospitalization (HFH) Rate at 1 Year Compared to the HF Hospitalization Rate in the Year Prior to Enrollment.
Description: HFH events at 1 year versus the HFH events in the year prior to enrollment
Time Frame: One year
Population: Patients who signed the Study Informed Consent and underwent successful CardioMEMS implant
Measure: Number (95% Confidence Interval); unit: HFH events per year
Arm/Group | Effectiveness Population
Number analyzed (Participants) | 299
HFH events per year
  Annualized HFH rate in the 12Months prior CardioMEMS implant | 1.59 [1.47 to 1.71]
  Annualized HFH rate in the 12Months post CardioMEMS implant | 0.49 [0.40 to 0.59]
  Annualized HFH rate post-Implant vs pre-implant | 0.31 [0.25 to 0.37]

ADVERSE EVENTS:
Time Frame: 2 years
Description: An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device under investigation.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 90/304
Serious Adverse Events (participants affected / at risk) | 225/304
Other Adverse Events (participants affected / at risk) | 17/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=304)
Abnormal heart rate or rhythm (Cardiac disorders) | 40 (54)
Allergic reaction (General disorders) | 1 (2)
Bleeding (Blood and lymphatic system disorders) | 3 (4)
Chest pain - cardiac (Cardiac disorders) | 14 (18)
Decompensated Heart Failure (Cardiac disorders) | 134 (267)
Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Myocardial Infarction (Cardiac disorders) | 4 (5)
Hematoma (Blood and lymphatic system disorders) | 2 (3)
Infection (Infections and infestations) | 43 (58)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 32 (37)
Sepsis (Infections and infestations) | 14 (15)
Thrombus (Vascular disorders) | 1 (1)
Transient ischemic attack (TIA) (Nervous system disorders) | 1 (1)
Valve Damage (Cardiac disorders) | 1 (1)
Other (General disorders) | 131 (212)
Hemoptisis (Vascular disorders) | 2 (2)
Lead dislodgement or migration (Product Issues) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=304)
Decompensated Heart Failure (Cardiac disorders) | 3 (3)
Infection (Infections and infestations) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (3)
Other (General disorders) | 7 (8)
Abnormal heart rate or rhythm (Cardiac disorders) | 1 (1)
Pulmonary infarct (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombus (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT02954341/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT02954341/ICF_001.pdf